CLINICAL TRIAL: NCT03481920
Title: A Pilot Trial of PEGPH20 (Pegylated Hyaluronidase) in Combination With Avelumab (Anti-PD-L1 MSB0010718C) in Chemotherapy Resistant Pancreatic Cancer
Brief Title: A Trial of PEGPH20 in Combination With Avelumab in Chemotherapy Resistant Pancreatic Cancer
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Stopped Enrollment
Sponsor: PH Research, S.L. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PH1603
Record Dates: First submitted 2018-02-10; First posted 2018-03-29 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-01

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Pancreatic Cancer
Keywords: pancreatic cancer, inmunotherapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — PEGPH20; avelumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PEGPH20 + Avelumab (Experimental): PEGPH20, a multi-site PEGylated enzyme generated by conjugating N-hydroxysuccinimidyl ester of methoxypoly(ethylene glycol)-butanoic acid (MSBA30K/B or PEG) and recombinant human hyaluronidase (rHuPH20). PEGPH20 has a half-life of approximately 2 days, thereby enabling systemic activity and sustained duration of action to degrade HA. In many different tumor types tested in murine xenograft models, response to PEGPH20 has been shown to be more robust for tumors characterized by higher HA expression.
  Interventions: Drug: PEGylated Recombinant Human Hyaluronidase (PEGPH20); Drug: Avelumab

INTERVENTIONS:
Drug: PEGylated Recombinant Human Hyaluronidase (PEGPH20) — PEGPH20 will be administered at a dose of 3.0 micrograms per kilogram (μg/kg) as an intravenous (IV) infusion.
Drug: Avelumab — Avelumab will be administered as at a dose of 10 milligrams per kilogram (mg/kg) as an intravenous (IV) infusion once every 2 weeks.
  Other Names: MSB0010718C

SUMMARY:
The purpose of this study is to evaluate the pharmacodynamics, safety and efficacy of PEGPH20 in combination with Avelumab in adult patients with chemotherapy resistant advanced or locally advanced pancreatic ductal adenocarcinoma (PDAC). This is a multi-center, open-label, non-randomized trial.

DETAILED DESCRIPTION:
The reported response rate with check-point inhibitors in PDAC is 0 %. This study tests the hypothesis that elimination of HA in pancreas tumor microenvironment mediated by PEG PH20 will result in increased tumor vascularization and vessel patency as well as stromal remodeling with increase immune infiltrate. These effects may facilitate the activity of check-point inhibitors like avelumab by at least two mechanisms including increase in drug delivery and increasing immune infiltrate.

The purpose of this study is to evaluate the pharmacodynamics, safety and efficacy of PEGPH20 in combination with Avelumab in adult patients with chemotherapy resistant advanced or locally advanced pancreatic ductal adenocarcinoma (PDAC). This is a multi-center, open-label, non-randomized trial.

ELIGIBILITY:
Key Inclusion Criteria:

* Signed, written IRB/IEC-approved Informed Consent Form
* Histologically or cytologically-confirmed pancreatic ductal adenocarcinoma (PDAC).
* Accessible tumor for two repeated tumor biopsies.
* Progression to first line treatment for locally advanced or advanced disease. Prior adjuvant chemotherapy or chemoradiation therapy for early disease is allowed.
* Age ≥18 years.
* Radiologically measurable disease per RECIST v1.1.
* Performance-status ECOG 0 -2.
* Life expectancy ≥ 3 months.
* Resolved acute effects of any prior therapy to baseline or Grade ≤1 severity
* Screening laboratory:

  1. Hematologic: ANC ≥ 1.5 × 109/L, platelet count ≥ 100 × 109/L, and hemoglobin ≥ 9 g/dL
  2. Hepatic: Total bilirubin level ≤ 1.5 × the ULN range and AST and ALT levels ≤ 2.5 × ULN or AST and ALT levels ≤ 5 X ULN (for subjects with documented metastatic disease to the liver)
  3. Renal: Estimated creatinine clearance ≥ 30 mL/min according to the Cockcroft-Gault formula or serum creatinine ≤ 2.0 mg/dL.
  4. Albumin ≥2.5 g/dL.
  5. Coagulation: PT time and INR within normal limits (+/-15%). PTT within normal limits (+/-15%).
* If a subject requires anticoagulation, treatment must be modified to enoxaparin.
* Negative serum pregnancy test if female subject is of childbearing potential.
* Patients who are willing and able to comply with scheduled visits, treatment plans, laboratory tests, biopsies when required, and other procedures.

Exclusion Criteria:

* Clinical evidence of DVT, PE, prior history of CVA or history of TIA within 12 months or other known TE event present during the screening period
* Current use of megestrol acetate (use within 10 days of Day 1).
* Contraindication to heparin as per institutional guidelines.
* Another primary cancer within the last 3 years currently requiring antineoplastic treatment within the exception of non-melanoma skin cancer, early-stage prostate cancer, or curatively treated cervical carcinoma in-situ.
* Current use of immunosuppressive medication within 2 weeks of study participation, EXCEPT for those listed in protocol
* Active autoimmune disease that might deteriorate when receiving an immuno-stimulatory agent: Patients with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment are eligible.
* Prior organ transplantation including allogenic stem-cell transplantation.
* Active infection requiring systemic therapy.
* Known infection with human immunodeficiency virus, Hepatitis B, or Hepatitis C
* Known prior severe hypersensitivity to investigational product, hyaluronidase, or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v4.03 Grade ≥ 3).
* Any history of anaphylaxis or uncontrolled asthma (that is, 3 or more features of partially controlled asthma).
* Clinically significant (i.e., active) cardiovascular disease: myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.
* Prior cerebrovascular accident/stroke.
* Clinically significant carotid artery disease (e.g. prior carotid surgery, symptomatic and/or requires treatment)
* Inability to comply with study and follow-up procedures as judged by the Investigator.
* Known alcohol or drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-06-10 (Actual)

PRIMARY OUTCOMES:
Determine ORR as per RECIST v1.1 criteria | 6 months from trial treatment initiation cycle 1/day 1. Each treatment cycle is 14 days
  Determine ORR as per RECIST v1.1 criteria
To assess the safety of this combination in patients with PDAC. | Initiation of trial treatment cycle 1/day 1 through 30 days after last dose of trial treatment
  graded by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03

SECONDARY OUTCOMES:
Determine OS (OVERALL SURVIVAL) | From date of treatment initiation cycle 1/day 1 until death from any cause, assessed up to 36 months
  The length of time from either the date of diagnosis or the start of treatment for a disease, such as cancer, that patients diagnosed with the disease are still alive
Determine PFS (PROGRESSION FREE SURVIVAL) | From date of treatment initiation cycle 1/day 1 until progression, assessed up to 24 months
  The length of time during and after the treatment of a disease, such as cancer, that a patient lives with the disease but it does not get worse.
Changes in CA 19,9 leves | Up to 4 weeks
  Measured in UI/ML

OTHER OUTCOMES:
The effect of PEGPH20 in tumor hyaluronic acid (HA) content in plasma and paired tumor biopsies of patients with PDAC treated with this regimen | tumor assessments performed every 8 +/- 1 week while on treatment, up to 24 months
  Hyaluronan concentrations will be analyzed in blood plasma samples by total HA disaccharides using liquid chromatography-tandem mass spectrometry (LC-MS-MS) . Hyaluronan concentrations will be analyzed in tumor tissue samples using an immunohistochemical method used exclusively in research.
Collagen content | tumor assessments performed every 8 +/- 1 week while on treatment, up to 24 months
  Collagen type I will be determine in tumor samples
Cancer associated fibroblasts (CAF) in tumor samples. | tumor assessments performed every 8 +/- 1 week while on treatment, up to 24 months
  Activated fibroblasts will be determined with double staining using vimentin as a fibroblast total marker and smooth muscle actin (SMA) as an activated fibroblast marker.
Immune infiltrate. | tumor assessments performed every 8 +/- 1 week while on treatment, up to 24 months
  CD4 and CD8 surface markers will be used to determine the immune infiltrate in tumor samples.

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Hospital Universitario Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Ramon y Cajal, Madrid